CLINICAL TRIAL: NCT04209192
Title: Randomized Phase II Study of Antibiotic Prophylaxis With Fosfomycin vs Amikacin in Transurethral Resection of Bladder
Brief Title: Antimicrobial Prophylaxis in Patients Who Underwent a Transurethral Resection of Bladder (TURB)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Laboratorios Senosiain, S.A. de C.V. (Industry)
Responsible Party: Principal Investigator, Ricardo Alonso Castillejos Molina, Urology Attending, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: URO-2995-19-20-1
Record Dates: First submitted 2019-12-18; First posted 2019-12-24 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Urinary Tract Infections; Bladder Cancer; Urologic Surgical Procedures
Keywords: UTI; Prophylaxis; Urinary Tract Infections; TURB; Fosfomycin; Amikacin; Transurethral Resection of Bladder
MeSH Terms: conditions — Urinary Tract Infections; Urinary Bladder Neoplasms | interventions — Fosfomycin; Amikacin

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Amikacin) (Active Comparator): Patients in the control group will receive amikacin as prophylactic antibiotic. It will be administered intravenously 30 minutes before procedure. Patients with an estimated glomerular filtration rate (EGFR) greater or equal than 70 ml/min will receive 1 gram of Amikacin. Patients with an EGFR less than 70 ml/min will received a calculated dose following the next parameters.
  Patients with EGFR between 69-40 ml/min should receive: the calculated GFR x 0.18 = mg/kg.
  Patients with EGFR less than 40 ml/min should receive: the calculated GFR x 0.36 = mg/kg.
  Interventions: Drug: Amikacin
- Intervention group (Fosfomycin) (Experimental): Patients in the intervention group will receive Fosfomycin trometamol as prophylactic antibiotic. It will be administered orally in the night before procedure. Patients must be on fasting and will receive 3 grams.
  Interventions: Drug: Fosfomycin Tromethamine 3G Sachet

INTERVENTIONS:
Drug: Fosfomycin Tromethamine 3G Sachet — Is the prophylactic drug which will be used in the intervention group.
  Other Names: Fosfomycin
  Arms: Intervention group (Fosfomycin)
Drug: Amikacin — Is the prophylactic drug which will be used in the control group.
  Other Names: Control
  Arms: Control group (Amikacin)

SUMMARY:
Antimicrobial prophylaxis in urological procedures is aimed to reduce the risk of local and systemic postoperative infections such as urinary tract infection or surgical site infection. It should be recommended only when the potential benefit exceeds the anticipated risks and costs. However, a wide variation in the use of periprocedural prophylactic antibiotics has been demonstrated, which frequently is incurred as an inappropriate selection of antimicrobials, inadequate schedule of administration or excessive duration of prophylaxis.

The increase in multidrug resistance of antibiotics in recent decades has been associated with its misuse, resulting in an increased rate of morbidity and mortality, prolonged hospital stays and increased care costs. Specifically, resistance to fluoroquinolones has increased its prevalence, a group of antibiotics widely used in urology. Therefore, local resistance patterns should be considered before following recommendations, especially in populations with poor control of antimicrobial use.

Transurethral resection of bladder (TURB) has become a frequent surgical procedure, as it is the main diagnostic and therapeutic tool for bladder cancer, representing the ninth most common malignancy in the world. However, no recent randomized clinical trial has investigated antimicrobial prophylaxis for TURB. It is well known that an expected complication of TURB is urinary tract infection (UTI), which is the most common healthcare related infection worldwide.

Under this premise, a randomized clinical trial is proposed to analyze the current panorama of UTI as a transcendent postoperative complication of TURB, under the context of the new emerging resistance parameters. The use of fosfomycin trometamol is proposed as a good potential option for urological procedures due to its high activity against multidrug-resistant gram-negative bacteria and its favorable pharmacokinetic parameters that guarantees wide tissue penetration and a high urinary concentration, in a single dose, the which will be compared with the control group with traditional prophylaxis (amikacin). The relative risk of UTI will be estimated, as well as the attributable risk of the main risk factors associated with this infection, allowing a better characterization of this population for adequate decision making regarding this clinical challenge.

DETAILED DESCRIPTION:
In 1931, Stern and McCarthy created the first practical cut-out resectoscope, allowing endoscopic diagnosis and treatment of bladder tumors for the first time in history. From now on, TURB has been the cornerstone of the management of bladder tumors. Histological evaluation is essential for the precise classification and staging of this cancer, as well as the therapeutic modality of choice for most patients with bladder cancer

Epidemiology Bladder cancer is the most common malignancy of the urinary tract, being the seventh most common cancer in men and number 17 in women. The worldwide incidence is 9 per 100,000 men and 2 per 100,000 women. More than 75,000 new cases of bladder cancer are diagnosed in the United States of America annually, making bladder cancer the ninth most common malignancy of the urinary tract. In addition, bladder cancer is responsible for 15,000 annual deaths in the United States of America, which makes it the thirteenth cause of death in general and the second most common cause of death among genitourinary tumors

In Latin America, bladder cancer has an incidence of 5.6 per 100,000 inhabitants. Mexico lacks reliable records of cancer epidemiology, however, in Mexico it corresponds to 14.4% of genitourinary cancers, ranking as the fourth most frequent. Mortality in men is 3 per 100,000 and in women 1 per 100,000 with very high geographical variation due to unequal access to health services. In a second level hospital in Mexico City were reported 861 cases of genitourinary cancer, bladder cancer was accounted for 13%.

Urinary tract infection as a postoperative complication In urology, the act of instrumentation is a potential contributor of infection risk.

Before finalizing the TURB, a urethral catheter is placed to irrigate and wash the bladder three times with 100 mL of saline. At the end of the procedure, the bladder is completely drained and the function of the catheter is guaranteed to assess a subsequent irrigation in the postoperative period, for complications that may occur, such as haematuria or urinary retention due to obstruction of a clot and / or irrigation of intravesical chemotherapy. In the absence of complications, the catheter can be removed after 24 hours.

The risk of urinary tract infection is directly proportional to the duration of the catheterization, measured in days (catheter days) and the surgical time. It is reported a mean catheter day of 1.9 +/- 1.7 in 130 post-TURB patients. It is well known that urinary tract infection (UTI) associated with catheter use is the most common healthcare related infection in the world and is the result of widespread use of urinary catheterization. The incidence reported of UTI in the literature after surgery is 5-10%. Antimicrobial prophylaxis in TURB decreases the risk of UTI from 10.1% to 2.9%. In a series of 10,559 patients in the United States of America the incidence of UTI in post-TURB patients was 3 to 5%, being the most observed complication. The investigators concluded that as surgery time increased, urinary tract infection increased (2.8% in 0-30min to 5.4% in> 90 min, P <0.001).

In addition, a patient with cancer is a host with increased susceptibility to acquire infections. In the last 50 years the epidemiology of bacterial infections in cancer patients has presented a continuous change influenced by the nature and intensity of chemotherapeutic and immunosuppressive regimes and the widespread use of empirical and prophylactic antibiotics

Antimicrobial prophylaxis in TURB Surgical antimicrobial prophylaxis is the systemic administration of an antibiotic before, during and / or shortly after a urological procedure aimed to reduce the risk of local and systemic postoperative infections, such as urinary tract infection or surgical site infection. The optimal antimicrobial drug should be a microbiologically active agent against the most frequent potential pathogens and must have good pharmacological properties.

Antibiotics The antibiotics used for prophylaxis must be effective against the characteristic bacterial microbiota of the surgical site and relevant to the disease. In addition, it must be considered the properties of the antimicrobial agent, such as cost, convenience and safety. It should reach tissue serum levels that exceed the minimum inhibitory concentration for microorganisms characteristic of the surgical site, in this case Enterobacteriaceae and Enterococci. Moreover, it must have a long half-life to maintain sufficient serum and tissue concentrations throughout the procedure without the need to administer another dose. It must be safe, cheap and unlikely to promote bacterial resistance.

For the urinary tract, cephalosporins, fluoroquinolones and aminoglycosides are generally effective, have a long half-life, are cheap (when used as a single dose) and are rarely associated with allergic reactions. In addition, fluoroquinolones and aminoglycosides can be used in patients with a beta-lactam allergy. These antimicrobials can effectively cover the expected organisms and meet the criteria indicated above.

Current recommendations and the context in Mexico The American Urological Association (AUA) and the Japanese guidelines recommend the use of fluoroquinolones, trimethoprim- sulfamethoxazole, penicillins, first or second generation cephalosporins or aminoglycosides before the start of TURB as an antimicrobial prophylaxis. According to the guidelines of the Canadian Urology Association (CUA), any randomized clinical trials of antimicrobial prophylaxis in TURB were found, so the recommendations about antibiotic prophylaxis are based on other endoscopic urological procedures. Use of fluoroquinolone are recommended for prophylaxis before surgical procedure, also trimethoprim- sulfamethoxazole or third generation cephalosporins can be used.

In a study of TURB in 2006, the investigators used oral levofloxacin 200mg as prophylactic antibiotic, which was given 30-60 minutes before the procedure. However, in this context it would not be convenient to use this regime, because in a study conducted in 2015 specified that countries with poor control of the use of antimicrobials such as Mexico, there is a trend towards bacterial resistance, placing fluoroquinolones as the second line of treatment in urinary tract infection . An important cause of the emergence of these resistant strains is the excessive use (treatment when it is not needed and prolonged exposure to therapy) of antimicrobial agents for all indications.

Fluoroquinolone-based regimens, a pillar of prophylaxis guidelines, are increasingly ineffective due to a constant increase in multidrug-resistant gram-negative bacteria (MDR). The same concerns apply with second and third generation cephalosporins, which have resistance problems and, if administered orally, do not have a good penetration in tissues such as prostate.

Problem definition Since 2000 a serious global public health problem has arisen in relation to the increase in antimicrobial resistance, particularly among the pathogens of the ESKAPE group (Enterococcus faecium, Staphylococcus aureus, Clostridium difficile, Acinetobacter species, Pseudomona aeruginosa and Enterobacteriaceae), which are microorganisms that cause urinary tract infection. In addition to the increase in multidrug resistance to antibiotics and their misuse, this has been associated with an increased rate of morbidity and mortality, prolonged hospital stay and increased care costs.That's why antimicrobial prophylaxis is of such magnitude and importance that it needs to be updated to its reasoned use in order to improve its performance.

In the case of TURB, there is little evidence in the literature that recommends the use of preoperative antimicrobial prophylaxis in TURB, due to the lack of studies on this subject. The incidence of UTI in TURB has been reported between 2 to 39% and risk of infection in TURB from 18 to 75%.

Justification Nosocomial infection has been associated with an increased length of postoperative stays, rate of hospital readmission and the outpatient use of antimicrobial agents, which significantly increases the costs and use of medical resources.

Optimally, the specific prophylactic regimen should be supported by clinical trials evidence. In many cases, randomized clinical trials are not available. Such lack of data does not impede the adequacy of some antibiotic regimes based on the efficacy of the drugs, the cost, safety and knowledge of the microbiota of the surgical site. When selecting the antimicrobial for prophylaxis, the clinician should be aware of the different resistance patterns in the local community. Specifically, resistance to fluoroquinolones, which has increased their prevalence, therefore, should be considered due to the high use of these agents for antimicrobial prophylaxis in urological surgery.

Regarding the premise, "surgical antimicrobial prophylaxis is recommended only when the potential benefit exceeds the risks and anticipated costs," information on the costs associated with the prophylactic use of antimicrobials specifically for urological surgery cannot be easily obtained, however, data from other surgical disciplines can guide us in making decisions. For example, the use of prophylaxis in transurethral resection of the prostate, where there are multiple clinical trials and it is recommended the use of prophylaxis with pre-procedure third-generation cephalosporins. On the contrary, excessive and / or inappropriate antimicrobial prophylaxis increases costs, which can be reduced with measures to improve commitment with evidence-based recommendations. In general, the financial costs of prophylaxis are controlled using the least expensive and safest effective agent for the shortest time that is compatible with good clinical practice.

There are currently few randomized clinical studies (conducted more than 25 years ago) on the subject. In 1988 a randomized clinical trial was conducted with 243 patients undergoing TURB, three perioperative doses of cefradine were compared with placebo, observing a significant reduction in the rate of bacteriuria. However, no similar randomized clinical trials have been performed, as well as for other cystoscopic procedures that involve transurethral manipulation (bladder biopsy, ureteral catheterization, laser prostatectomy, etc.). For this reason, updated and available evidence is required for this widely used procedure.

The American Urological Association and the Japanese guidelines recommend the use of fluoroquinolones, trimethoprim, penicillins, first or second generation cephalosporins or aminoglycosides before the start of TURB as an antimicrobial prophylaxis In countries with poor control of the use of antimicrobials such as Mexico, there is a tendency towards bacterial resistance, placing fluoroquinolones as the second line of treatment for urinary tract infection. Therefore, the use of fluoroquinolone-based regimens, a pillar of prophylaxis guidelines, is increasingly ineffective due to a constant increase in resistant multidrug gram negative bacteria. The same applies with second and third generation cephalosporins, which also have resistance problems.

In 2007 a randomized clinical trial was performed and the effectiveness of fosfomycin against cefotiam to prevent infections associated with urological surgery was compared ,the response rates reported were 92.9% for fosfomycin and 94.9% for cefotiam in patients with transurethral surgery. Therefore, fosfomycin trometamol may be a potential option for urological procedures, due to its high effectiveness against resistant multidrug gram negative bacteria and its favorable pharmacokinetic parameters.

The aim of the study is to provide evidence to help clarify the usefulness and feasibility of antimicrobial prophylaxis, being fosfomycin trometamol an antibiotic that meets the necessary characteristics for this intervention. Therefore it will contribute to the characterization of the population that undergoes this procedure, which includes the description of risk factors and microbiological characteristics, such as the identification of emerging resistant strains. The results obtained will contribute towards the decision-making of this and other cytoscopic procedures due to the similarities in terms of invasiveness and possible tissue trauma, suggesting that the data regarding transurethral bladder resection can reasonably be extrapolated to other cystoscopic procedures with manipulation. The above will be compared with the antimicrobial prophylaxis that usually occurs in the Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran which is based on aminoglycosides (Amikacin) administered in anesthetic induction before the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old of age
* Patients with a programmed TURB
* Absence of urinary tract infection (negative urine culture and no clinical manifestations for urinary tract infection)

Exclusion Criteria:

* Patients with asymptomatic bacteriuria
* Patients with positive urine culture before procedure
* Patients with urinary catheterization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence of urinary tract infection after transurethral resection of bladder | 30 days after procedure
  Measurement tool: Clinical manifestations of urinary tract infection plus positive urine culture.
  Measurement unit: Colony-forming unit (CFU) per milliliter (mL) depending on how the urine sample was took. A positive urine culture will be confirmed using the next parameters: For midstream urine a count greater or equal to 100,000 CFU/mL and for urine obtained from a urethral catheter a count a count greater or equal to 100 CFU/mL Clinical manifestations of urinary tract infection: Patient presenting 1 or more of the following signs or symptoms: fever, dysuria, frequency, hematuria, lumbar pain, costovertebral angle tenderness)
Incidence of asymptomatic bacteriuria after transurethral resection of bladder | 30 days after procedure
  Measurement tool: Positive urine culture and no clinical manifestation of urinary tract infection Measurement unit: Colony-forming unit (CFU) per milliliter (mL) depending on how the urine sample was took. A urine culture will be positive using the next parameters: For midstream urine a count greater or equal to 100,000 CFU/mL and for urine obtained from a urethral catheter a count a count greater or equal to 100 CFU/mL No clinical manifestations of urinary tract infection
Relative risk of asymptomatic bacteriuria after transurethral resection of bladder | 30 days after procedure
  Measurement tool: Positive urine culture and no clinical manifestation of urinary tract infection Measurement unit: Colony-forming unit (CFU) per milliliter (mL) depending on how the urine sample was took. A urine culture will be positive using the next parameters: For midstream urine a count greater or equal to 100,000 CFU/mL and for urine obtained from a urethral catheter a count a count greater or equal to 100 CFU/mL No clinical manifestations of urinary tract infection
Relative Risk of urinary tract infection after transurethral resection of bladder | 30 days after procedure
  Measurement tool: Clinical manifestations of urinary tract infection plus positive urine culture.
  Measurement unit: Colony-forming unit (CFU) per milliliter (mL) depending on how the urine sample was took. A positive urine culture will be confirmed using the next parameters: For midstream urine a count greater or equal to 100,000 CFU/mL and for urine obtained from a urethral catheter a count a count greater or equal to 100 CFU/mL Clinical manifestations of urinary tract infection: Patient presenting 1 or more of the following signs or symptoms: fever, dysuria, frequency, hematuria, lumbar pain, costovertebral angle tenderness)

SECONDARY OUTCOMES:
Relative risk of patients presenting a single bladder tumor | During procedure
  Measurement tool: Observation of the procedure and report of data collection sheet Measurement unit: Patients that presented a single tumor: positive Patients presenting more than 1 tumor: negative
% of patients presenting a single bladder tumor | During procedure
  Measurement tool: Observation of the procedure and report of data collection sheet Measurement unit: Patients that presented a single tumor: positive Patients presenting more than 1 tumor: negative
Relative risk of patients presenting 2 to 7 bladder tumors | During procedure
  Measurement tool: Observation of the procedure and report of data collection sheet Measurement unit: Patients that presented 2 to 7 tumors: positive Patients that presented more than 7 tumors or a single tumor: negative
% of patients presenting 2 to 7 bladder tumors | During procedure
  Measurement tool: Observation of the procedure and report of data collection sheet Measurement unit: Patients that presented 2 to 7 tumors: positive Patients that presented more than 7 tumors or a single tumor: negative
Relative risk of patients presenting more than 7 bladder tumors | During procedure
  Measurement tool: Observation of the procedure and report of data collection sheet Measurement unit: Patients that presented more than 7 tumors: positive Patients that presented less than 8 tumors: negative
% of patients presenting more than 7 bladder tumors | During procedure
  Measurement tool: Observation of the procedure and report of data collection sheet Measurement unit: Patients that presented more than 7 tumors: positive Patients that presented less than 8 tumors: negative
Relative risk of bleeding during surgery | During procedure
  Measurement tool: Observation of the procedure and report of data collection sheet Measurement unit: milliliters
Relative risk of patients with I on ASA classification | During procedure
  Measurement tool: Observation of the procedure and report of data collection sheet Measurement unit: Patient with I ASA classification: Positive Patient with other ASA classification not being I: Negative
% of patients with I on ASA classification | During procedure
  Measurement tool: Observation of the procedure and report of data collection sheet Measurement unit: Patient with I ASA classification: Positive Patient with other ASA classification not being I: Negative
Relative risk of patients with II on ASA classification | During procedure
  Measurement tool: Observation of the procedure and report of data collection sheet Measurement unit: Patient with II ASA classification: Positive Patient with other ASA classification not being II: Negative
% of patients with II on ASA classification | During procedure
  Measurement tool: Observation of the procedure and report of data collection sheet Measurement unit: Patient with II ASA classification: Positive Patient with other ASA classification not being II: Negative
Relative risk of patients with III on ASA classification | During procedure
  Measurement tool: Observation of the procedure and report of data collection sheet Measurement unit: Patient with III ASA classification: Positive Patient with other ASA classification not being III: Negative
% of patients with III on ASA classification | During procedure
  Measurement tool: Observation of the procedure and report of data collection sheet Measurement unit: Patient with III ASA classification: Positive Patient with other ASA classification not being III: Negative
Relative risk of patients with IV on ASA classification | During procedure
  Measurement tool: Observation of the procedure and report of data collection sheet Measurement unit: Patient with IV ASA classification: Positive Patient with other ASA classification not being IV: Negative
% of patients with IV on ASA classification | During procedure
  Measurement tool: Observation of the procedure and report of data collection sheet Measurement unit: Patient with IV ASA classification: Positive Patient with other ASA classification not being IV: Negative
Relative risk of patients with a urethral catheter removed 24 hours after procedure | 1 day after procedure
  Measurement tool: Observation of the procedure, report of data collection sheet and follow up note review Measurement unit: Patient with a urethral catheter removed 24 hours after procedure: positive Patient with a urethral catheter after 24 hours after procedure: negative
% of patients with a urethral catheter removed 24 hours after procedure | 1 day after procedure
  Measurement tool: Observation of the procedure, report of data collection sheet and follow up note review Measurement unit: Patient with a urethral catheter removed 24 hours after procedure: positive Patient with a urethral catheter after 24 hours after procedure: negative
Relative risk of muscle invasive bladder cancer | 30 days after procedure
  Based on the results of the histopathology report, the patients will be classified in nominal groups (non-muscle invasive bladder tumor, muscle invasive bladder tumor, chronic cystitis or other)
  Measurement tool: Histopathology report Measurement unit: Patient with muscle invasive bladder cancer: Positive Patient with non-muscle invasive bladder cancer or chronic cystitis: Negative
% of patients with muscle invasive bladder cancer | 30 days after procedure
  Based on the results of the histopathology report, the patients will be classified in nominal groups (non-muscle invasive bladder tumor, muscle invasive bladder tumor, chronic cystitis or other) Measurement tool: Histopathology report Measurement unit: Patient with muscle invasive bladder cancer: Positive Patient with non-muscle invasive bladder cancer or chronic cystitis: Negative
Relative risk of non-muscle invasive bladder cancer | 30 days after procedure
  Based on the results of the histopathology report, the patients will be classified in nominal groups (non-muscle invasive bladder tumor, muscle invasive bladder tumor, chronic cystitis or other) Measurement tool: Histopathology report Measurement unit: Patient with non-muscle invasive cancer: Positive Patient with muscle invasive cancer or chronic cystitis: Negative
% of patients with non-muscle invasive bladder cancer | 30 days after procedure
  Based on the results of the histopathology report, the patients will be classified in nominal groups (non-muscle invasive bladder tumor, muscle invasive bladder tumor, chronic cystitis or other) Measurement tool: Histopathology report Measurement unit: Patient with non-muscle invasive bladder cancer: Positive Patient with muscle invasive bladder cancer or chronic cystitis: Negative
Relative risk of chronic cystitis | 30 days after procedure
  Based on the results of the histopathology report, the patients will be classified in nominal groups (non-muscle invasive bladder tumor, muscle invasive bladder tumor, chronic cystitis or other) Measurement tool: Histopathology report Measurement unit: Patient with chronic cystitis: Positive Patient with non-muscle invasive bladder cancer or muscle invasive bladder cancer: Negative
% of patients with chronic cystitis | 30 days after procedure
  Based on the results of the histopathology report, the patients will be classified in nominal groups (non-muscle invasive bladder tumor, muscle invasive bladder tumor, chronic cystitis or other) Measurement tool: Histopathology report Measurement unit: Patient with chronic cystitis: Positive Patient with non-muscle invasive bladder cancer or muscle invasive bladder cancer: Negative
Relative risk of number of days of urethral catheter after procedure | 30 days after procedure
  Measurement tool: Observation of the procedure, report of data collection sheet and follow up note review Measurement unit: Number of days of urethral catheter after procedure

OTHER OUTCOMES:
Relative risk of positive nitrites in preoperative urinalysis | 30 days before procedure
  Measurement tool: Urinalysis Measurement unit: Presence of nitrites in urinalysis: positive. Absence of nitrites in urinalysis: negative
Relative risk of positive leukocytes in urine in preoperative urinalysis | 30 days before procedure
  Measurement tool: Urinalysis and microscopy Measurement unit: Presence of 0-5 leukocytes per field in urinalysis: negative.
  Presence of 6 or more leukocytes per field in urinalysis: positive
Relative risk of positive erythrocytes in urine in preoperative urinalysis | 30 days before procedure
  Measurement tool: Urinalysis and microscopy Measurement unit: Presence of 0-2 erythrocytes per field in urinalysis: negative.
  Presence of 3 or more erythrocytes per field in urinalysis: positive
Relative risk of antibiotic use in the past 3 months | 15 days before procedure
  Measurement tool: Interrogation and questionnaire Measurement unit: Use of antibiotics in the past 3 months before procedure: positive.
  No use of antibiotics in the past 3 months before procedure: negative.
% of patients that used antibiotics in the past 3 months | 15 days before procedure
  Measurement tool: Interrogation and questionnaire Measurement unit: Use of antibiotics in the past 3 months before procedure: positive.
  No use of antibiotics in the past 3 months before procedure: negative.
Relative risk of patients that had a urinary tract infection before procedure | 15 days before procedure
  Measurement tool: Interrogation, questionnaire and clinical file review. Measurement unit: Number of times the patient had a urinary tract infection before procedure.
% of patients that had an urinary tract infection before procedure | 15 days before procedure
  Measurement tool: Interrogation, questionnaire and clinical file review. Measurement unit: Number of times the patient had a urinary tract infection before procedure.
Relative risk of patients that had a urological surgery before procedure | 15 days before procedure
  Measurement tool: Interrogation, questionnaire and clinical file review. Measurement unit: Patients had a urological surgery before procedure: positive Patient did not had a urological surgery before procedure: negative
% of patients that had a urological surgery before procedure | 15 days before procedure
  Measurement tool: Interrogation, questionnaire and clinical file review. Measurement unit: Patients had a urological surgery before procedure: positive Patient did not had a urological surgery before procedure: negative
Relative risk of patients that had a cystoscopy before procedure | 15 days before procedure
  Measurement tool: Interrogation, questionnaire and clinical file review. Measurement unit: Patient had cystoscopy before procedure: positive Patient did not had a cystoscopy before procedure: negative
% of patients that had a cystoscopy before procedure | 15 days before procedure
  Measurement tool: Interrogation, questionnaire and clinical file review. Measurement unit: Patient had cystoscopy before procedure: positive Patient did not had a cystoscopy before procedure: negative
Relative risk of patients that have a urinary malformation before procedure | 15 days before procedure
  Measurement tool: Interrogation, questionnaire and clinical file review. Measurement unit: Patient had urinary malformation before procedure: positive Patient did not had a urinary malformation before procedure: negative
% of patients that have a urinary malformation before procedure | 15 days before procedure
  Measurement tool: Interrogation, questionnaire and clinical file review. Measurement unit: Patient had urinary malformation before procedure: positive Patient did not had a urinary malformation before procedure: negative
Relative risk of patients that had obstructive uropathy before procedure | 15 days before procedure
  Measurement tool: Interrogation, questionnaire and clinical file review. Measurement unit: Patient had obstructive uropathy before procedure: positive Patient did not had a obstructive uropathy before procedure: negative
% of patients that had obstructive uropathy before procedure | 15 days before procedure
  Measurement tool: Interrogation, questionnaire and clinical file review. Measurement unit: Patient had obstructive uropathy before procedure: positive Patient did not had a obstructive uropathy before procedure: negative
Relative risk of patients that had vesicoureteral reflux before procedure | 15 days before procedure
  Measurement tool: Interrogation, questionnaire and clinical file review. Measurement unit: Patient had vesicoureteral reflux before procedure: positive Patient did not had vesicoureteral reflux before procedure: negative
% of patients that had vesicoureteral reflux before procedure | 15 days before procedure
  Measurement tool: Interrogation, questionnaire and clinical file review. Measurement unit: Patient had vesicoureteral reflux before procedure: positive Patient did not had vesicoureteral reflux before procedure: negative
Relative risk of patients that had a transurethral resection of bladder before procedure | 15 days before procedure
  Measurement tool: Interrogation, questionnaire and clinical file review. Measurement unit: Number of times the patient had a transurethral resection of bladder tumor before procedure
% patients that did not had a transurethral resection of bladder before procedure | 15 days before procedure
  Measurement tool: Interrogation, questionnaire and clinical file review. Measurement unit: Number of times the patient had a transurethral resection of bladder tumor before procedure
Relative risk of patients who received intravesical chemotherapy before procedure | 15 days before procedure
  Measurement tool: Interrogation and questionnaire Measurement unit: Use of intravesical chemotherapy before procedure: positive. Use of intravesical chemotherapy before procedure: negative.
% of patients who received intravesical chemotherapy before procedure | 15 days before procedure
  Measurement tool: Interrogation and questionnaire Measurement unit: Use of intravesical chemotherapy before procedure: positive. Patient did not had intravesical chemotherapy before procedure: negative.
Relative risk of patients who received intravesical immunotherapy with BCG before procedure | 15 days before procedure
  Measurement tool: Interrogation and questionnaire Measurement unit: Use of intravesical immunotherapy with BCG before procedure: positive.
  Patient did not had intravesical immunotherapy with BCG before procedure: negative.
% of patients who received intravesical immunotherapy with BCG before procedure | 15 days before procedure
  Measurement tool: Interrogation and questionnaire Measurement unit: Use of intravesical immunotherapy with BCG before procedure: positive.
  Patient did not had intravesical immunotherapy with BCG before procedure: negative.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Castillejos, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herr HW, Donat SM, Reuter VE. Management of low grade papillary bladder tumors. J Urol. 2007 Oct;178(4 Pt 1):1201-5; discussion 1205. doi: 10.1016/j.juro.2007.05.148. Epub 2007 Aug 14. PMID 17698090
- [Background] Holzbeierlein JM, Smith JA Jr. Surgical management of noninvasive bladder cancer (stages Ta/T1/CIS). Urol Clin North Am. 2000 Feb;27(1):15-24, vii-viii. doi: 10.1016/s0094-0143(05)70230-5. PMID 10696241
- [Background] Mayorga, G; Ibarra, O; Sedano, B; Trujillo, O; Cornejo, D; Palmeros, R;…Pacheco, G. (2014) Aplicación de nomogramas en México para cáncer de vejiga en pacientes del Hospital General "Dr Manuel Gea González". Revista Mexicana de Urología, 74(1),3-8. https://doi.org/10.1016/s2007-4085(15)30002-1
- [Background] Parkin DM. The global burden of urinary bladder cancer. Scand J Urol Nephrol Suppl. 2008 Sep;(218):12-20. doi: 10.1080/03008880802285032. PMID 19054893
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Sedano-Basilio, J; Mayorga-Gómez, E; Garza-Sainz, G; Conrejo-Dávila, V; Uberetagoyena-Tello de Meneses, I; Palmeros-Rodríguez, A;… Pacheco-Gahbler, C. (2016) Epidemiología de los tumores genitourinarios en una década. Revista Mexicana de Urología, 76(3), 131-140. https://doi.org/10.1016/j.uromx.2016.01.004
- [Background] Pycha, A. & Palermo, S. (2005) Transurethral Resection of Bladder Tumors. In R. Hoenfellner & J. Stolzenburg (Eds.) Manual Endourology (pp. 55-70) Berlín: Springer
- [Background] Hooton TM, Bradley SF, Cardenas DD, Colgan R, Geerlings SE, Rice JC, Saint S, Schaeffer AJ, Tambayh PA, Tenke P, Nicolle LE; Infectious Diseases Society of America. Diagnosis, prevention, and treatment of catheter-associated urinary tract infection in adults: 2009 International Clinical Practice Guidelines from the Infectious Diseases Society of America. Clin Infect Dis. 2010 Mar 1;50(5):625-63. doi: 10.1086/650482. PMID 20175247
- [Background] Junuzovic D, Hasanbegovic M, Zvizdic S, Hamzic S, Zunic L. The connection between endourological procedures and occurrence of urinary infections. Mater Sociomed. 2014 Aug;26(4):237-41. doi: 10.5455/msm.2014.237-241. Epub 2014 Aug 26. PMID 25395884
- [Background] Alsaywid BS, Smith GH. Antibiotic prophylaxis for transurethral urological surgeries: Systematic review. Urol Ann. 2013 Apr;5(2):61-74. doi: 10.4103/0974-7796.109993. PMID 23798859
- [Background] Matulewicz RS, Sharma V, McGuire BB, Oberlin DT, Perry KT, Nadler RB. The effect of surgical duration of transurethral resection of bladder tumors on postoperative complications: An analysis of ACS NSQIP data. Urol Oncol. 2015 Aug;33(8):338.e19-24. doi: 10.1016/j.urolonc.2015.05.011. Epub 2015 Jun 10. PMID 26072111
- [Background] Rolston K.V. (2003) Pseudomonas Aeruginosa Infections in Cancer Patients. In: Hauser A.R., Rello J. (eds) Severe Infections Caused by Pseudomonas Aeruginosa. Perspectives on Critical Care Infectious Diseases, vol 7. Springer, Boston, MA
- [Background] Mazzei T, Diacciati S. Pharmacological aspects of the antibiotics used for urological diagnostic procedures. J Chemother. 2014 Oct;26 Suppl 1:S24-34. doi: 10.1179/1120009X14Z.000000000234. PMID 25245708
- [Background] Wolf JS Jr, Bennett CJ, Dmochowski RR, Hollenbeck BK, Pearle MS, Schaeffer AJ; Urologic Surgery Antimicrobial Prophylaxis Best Practice Policy Panel. Best practice policy statement on urologic surgery antimicrobial prophylaxis. J Urol. 2008 Apr;179(4):1379-90. doi: 10.1016/j.juro.2008.01.068. Epub 2008 Feb 20. PMID 18280509
- [Background] Yamamoto S, Shigemura K, Kiyota H, Wada K, Hayami H, Yasuda M, Takahashi S, Ishikawa K, Hamasuna R, Arakawa S, Matsumoto T; Japanese Research Group for UTI. Essential Japanese guidelines for the prevention of perioperative infections in the urological field: 2015 edition. Int J Urol. 2016 Oct;23(10):814-824. doi: 10.1111/iju.13161. Epub 2016 Aug 16. PMID 27531443
- [Background] Mrkobrada M, Ying I, Mokrycke S, Dresser G, Elsayed S, Bathini V, Boyce E, Luke P. CUA Guidelines on antibiotic prophylaxis for urologic procedures. Can Urol Assoc J. 2015 Jan-Feb;9(1-2):13-22. doi: 10.5489/cuaj.2382. No abstract available. PMID 25737749
- [Background] Yokoyama M, Fujii Y, Yoshida S, Saito K, Koga F, Masuda H, Kobayashi T, Kawakami S, Kihara K. Discarding antimicrobial prophylaxis for transurethral resection of bladder tumor: a feasibility study. Int J Urol. 2009 Jan;16(1):61-3. doi: 10.1111/j.1442-2042.2008.02188.x. PMID 19120528
- [Background] Sotomayor-de Zavaleta, M; Ponce de León-Garduño, A; Guzmán-Esquivel, J. & Rosas-Nava, E. (2015). Recomendaciones de expertos mexicanos en en tratamiento de las infecciones del tracto urinario en pacientes adultos, embarazadas y niños. Revista Mexicana de Urología, 72 (2), 1-46
- [Background] Boucher HW, Talbot GH, Bradley JS, Edwards JE, Gilbert D, Rice LB, Scheld M, Spellberg B, Bartlett J. Bad bugs, no drugs: no ESKAPE! An update from the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jan 1;48(1):1-12. doi: 10.1086/595011. PMID 19035777
- [Background] Panach-Navarrete J, Valls-Gonzalez L, Sanchez-Cano E, Medina-Gonzalez M, Castello-Porcar A, Martinez-Jabaloyas JM. Comparison of three different antibiotic protocols in transurethral resection of bladder tumour and the possible infectious risk factors: A non-randomized, prospective study. Can Urol Assoc J. 2018 Nov;12(11):E466-E674. doi: 10.5489/cuaj.5207. Epub 2018 Jun 8. PMID 29989880
- [Background] Junuzovic, D; Hasanbegovic, M. & Kovacevic-Prstojevic, J (2011) The Incidence of Acquired Urinary Tract Infections in patients After Transurethral Resection of Bladder Tumors. MSM, 23 (2): 91-92
- [Background] Herwaldt LA, Cullen JJ, Scholz D, French P, Zimmerman MB, Pfaller MA, Wenzel RP, Perl TM. A prospective study of outcomes, healthcare resource utilization, and costs associated with postoperative nosocomial infections. Infect Control Hosp Epidemiol. 2006 Dec;27(12):1291-8. doi: 10.1086/509827. Epub 2006 Nov 17. PMID 17152025
- [Background] Andriole VT. The quinolones: past, present, and future. Clin Infect Dis. 2005 Jul 15;41 Suppl 2:S113-9. doi: 10.1086/428051. PMID 15942877
- [Background] Delavierre D, Huiban B, Fournier G, Le Gall G, Tande D, Mangin P. [The value of antibiotic prophylaxis in transurethral resection of bladder tumors. Apropos of 61 cases]. Prog Urol. 1993 Aug-Sep;3(4):577-82. French. PMID 8401618
- [Background] Upton JD, Das S. Prophylactic antibiotics in transurethral resection of bladder tumors: are they necessary? Urology. 1986 May;27(5):421-3. doi: 10.1016/0090-4295(86)90406-1. PMID 3518183
- [Background] MacDermott JP, Ewing RE, Somerville JF, Gray BK. Cephradine prophylaxis in transurethral procedures for carcinoma of the bladder. Br J Urol. 1988 Aug;62(2):136-9. doi: 10.1111/j.1464-410x.1988.tb04292.x. PMID 3044484
- [Background] Ishizaka K, Kobayashi S, Machida T, Yoshida K. Randomized prospective comparison of fosfomycin and cefotiam for prevention of postoperative infection following urological surgery. J Infect Chemother. 2007 Oct;13(5):324-31. doi: 10.1007/s10156-007-0544-5. Epub 2007 Oct 30. PMID 17982722
- [Background] Patel SS, Balfour JA, Bryson HM. Fosfomycin tromethamine. A review of its antibacterial activity, pharmacokinetic properties and therapeutic efficacy as a single-dose oral treatment for acute uncomplicated lower urinary tract infections. Drugs. 1997 Apr;53(4):637-56. doi: 10.2165/00003495-199753040-00007. PMID 9098664